CLINICAL TRIAL: NCT01510002
Title: Prophylactic Central Neck Dissection for Papillary Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Marcin Barczynski, Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BBN/501/ZKL/1447
Record Dates: First submitted 2012-01-09; First posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Papillary Thyroid Cancer
Keywords: papillary thyroid cancer; central neck dissection; survival; locoregional control; morbidity
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TT (Active Comparator): Extracapsular total thyroidectomy
  Interventions: Procedure: Total thyroidectomy
- TT+CND (Experimental): Extracapsular total thyroidectomy puls prophylactic central neck dissection
  Interventions: Procedure: Total thyroidectomy + prophylactic central neck dissection

INTERVENTIONS:
Procedure: Total thyroidectomy — Extracapsular total thyroidectomy
  Arms: TT
Procedure: Total thyroidectomy + prophylactic central neck dissection — Extracapsular total thyroidectomy plus prophylactic central neck dissection
  Arms: TT+CND

SUMMARY:
The purpose of this study is to determine whether prophylactic central neck dissection is beneficial for patients with papillary thyroid cancer staged preoperatively as node negative.

DETAILED DESCRIPTION:
Several respected organizations have recently recommended that total thyroidectomy plus prophylactic central neck dissection should be the standard operation for papillary thyroid cancer. However, it is still unclear if this approach has any benefit on survival or locoregional control of the disease. In addition, potential advantages of this more aggressive surgical approach should outweigh the risk of morbidity. The purpose of this retrospective cohort study is to determine whether prophylactic central neck dissection is beneficial for patients with papillary thyroid cancer staged preoperatively as node negative. In this study outcomes of total thyroidectomy versus this plus prophylactic central neck dissection for papillary thyroid cancer are compared in a 10-year follow-up. Patients operated between 1993 and 1997 (n=282) underwent total thyroidectomy alone, whereas patients operated between 1998 and 2002 (n=358) underwent total thyroidectomy plus prophylactic central neck dissection.

ELIGIBILITY:
Inclusion Criteria:

* a pathological diagnosis of papillary thyroid cancer,
* in a patient with negative cervical lymph nodes on pre-, or intraoperative evaluation

Exclusion Criteria:

* incidental diagnosis of papillary thyroid cancer following hemithyroidectomy and requiring completion thyroidectomy,
* one-stage lymph nodes dissection based on therapeutic intent,
* previous thyroid surgery,
* incomplete follow-up information,
* incomplete histopathology report,
* ASA grade higher than 3 (American Society of Anesthesiology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 1993-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 10 years
disease-specific survival | up to 10 years
locoregional control | up to 10 years

SECONDARY OUTCOMES:
number of patients with negative serum thyroglobulin levels | up to 10 years
postoperative morbidity rate (hypoparathyroidism and recurrent laryngeal nerve injury). | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczynski, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian Univerity, Medical College, 3rd Department of General Surgery, Krakow, Malopolska, Poland

REFERENCES:
- [Background] Forest VI, Clark JR, Ebrahimi A, Cho EA, Sneddon L, Gao K, O'brien CJ. Central compartment dissection in thyroid papillary carcinoma. Ann Surg. 2011 Jan;253(1):123-30. doi: 10.1097/SLA.0b013e3181fc9644. PMID 21135696
- [Background] Mulla M, Schulte KM. Central cervical lymph node metastases in papillary thyroid cancer: a systematic review of imaging-guided and prophylactic removal of the central compartment. Clin Endocrinol (Oxf). 2012 Jan;76(1):131-6. doi: 10.1111/j.1365-2265.2011.04162.x. PMID 21722150
- [Background] Popadich A, Levin O, Lee JC, Smooke-Praw S, Ro K, Fazel M, Arora A, Tolley NS, Palazzo F, Learoyd DL, Sidhu S, Delbridge L, Sywak M, Yeh MW. A multicenter cohort study of total thyroidectomy and routine central lymph node dissection for cN0 papillary thyroid cancer. Surgery. 2011 Dec;150(6):1048-57. doi: 10.1016/j.surg.2011.09.003. PMID 22136820
- [Background] Alvarado R, Sywak MS, Delbridge L, Sidhu SB. Central lymph node dissection as a secondary procedure for papillary thyroid cancer: Is there added morbidity? Surgery. 2009 May;145(5):514-8. doi: 10.1016/j.surg.2009.01.013. Epub 2009 Mar 27. PMID 19375610
- [Background] Grodski S, Cornford L, Sywak M, Sidhu S, Delbridge L. Routine level VI lymph node dissection for papillary thyroid cancer: surgical technique. ANZ J Surg. 2007 Apr;77(4):203-8. doi: 10.1111/j.1445-2197.2007.04019.x. PMID 17388820
- [Background] Moo TA, Umunna B, Kato M, Butriago D, Kundel A, Lee JA, Zarnegar R, Fahey TJ 3rd. Ipsilateral versus bilateral central neck lymph node dissection in papillary thyroid carcinoma. Ann Surg. 2009 Sep;250(3):403-8. doi: 10.1097/SLA.0b013e3181b3adab. PMID 19661784
- [Background] Barczynski M, Konturek A, Stopa M, Cichon S, Richter P, Nowak W. Total thyroidectomy for benign thyroid disease: is it really worthwhile? Ann Surg. 2011 Nov;254(5):724-29; discussion 729-30. doi: 10.1097/SLA.0b013e3182360118. PMID 22005150
- [Derived] Barczynski M, Konturek A, Stopa M, Nowak W. Prophylactic central neck dissection for papillary thyroid cancer. Br J Surg. 2013 Feb;100(3):410-8. doi: 10.1002/bjs.8985. Epub 2012 Nov 27. PMID 23188784